CLINICAL TRIAL: NCT06507514
Title: Safety and Efficacy of Blinatumomab and Autologous HSCT Sandwich Strategy as Consolidation Therapy for B-cell Acute Lymphoblastic Leukemia
Brief Title: Blinatumomab and Auto-HSCT Sandwich Strategy as Consolidation Therapy for B-ALL
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Sheng-Li Xue, MD, professor, The First Affiliated Hospital of Soochow University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SZBALL02
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: B-cell Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma | interventions — blinatumomab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blinatumomab and Auto-HSCT Sandwich Strateg (Other)
  Interventions: Combination Product: blinatumomab and auto-HSCT "sandwich " strategy

INTERVENTIONS:
Combination Product: blinatumomab and auto-HSCT "sandwich " strategy — The patients received sequential infusion of blinatumomab after standard induction and consolidation chemotherapy. Autologous stem cells mobilization and collection were performed 6-8 weeks after infusion. Following successful stem cell collection, autologous stem cell transplantation was conducted. Starting from the third month after autologous stem cell transplantation, the second maintenance treatment with brentuximab vedotin was administered, with one cycle every three months, for a total of four cycles. Patients were followed up and minimal residual diseases (MRD) was monitored by flow cytometry and second-generation gene sequencing of IgH rearrangement.

SUMMARY:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is the main method potentially curing adult B-ALL, but the high treatment-related mortality (NRM) affects overall survival (OS). Autologous stem cell transplantation (auto-HSCT) can significantly reduce NRM but has a higher relapse rate. Studies have confirmed that achieving MRD negativity before Auto-HSCT can effectively reduce post-transplant relapse, achieving similar efficacy to allo-HSCT. The efficacy of blinatumomab in clearing MRD has been confirmed. Therefore, using blinatumomab combined with Auto-HSCT for B-ALL patients seems to make it possible to achieve benefits in leukemia free survival（LFS） and OS. The investigators first conducted blinatumomab and auto-HSCT "sandwich " strategy as consolidation therapy in patients with B-ALL. The main Purpose of this study was to observe the safety and efficacy of this new strategy.

DETAILED DESCRIPTION:
Enrolled patients received induction chemotherapy with the IVP regimen and two cycles of consolidation chemotherapy: high-dose cytarabine (Ara-c) + pegaspargase (± Tyrosine kinase inhibitors ,TKI) and methotrexate (MTX) + pegaspargase (± TKI). Sequential treatment with blinatumomab was then administered. After the first treatment with blinatumomab, autologous stem cell mobilization and collection were performed. Following successful stem cell collection, autologous stem cell transplantation was conducted. Starting from the third month after autologous stem cell transplantation, the second maintenance treatment with blinatumomab was administered, with one cycle every three months, for a total of four cycles. Long-term follow-up monitoring was then conducted. The follow-up period for this study was two years, and data on two-year LFS, OS, and NRM rates were collected.

ELIGIBILITY:
Inclusion Criteria:

* subjects with a primary diagnosis of B-ALL who have any of the following: (a) no suitable allogeneic HSCT donor. (b) refusal of allogeneic HSCT.
* positive expression of CD19 in peripheral blood or bone marrow primary cells detected by flow cytometry.
* ardiac ultrasound left ventricular ejection fraction ≥ 50%; Creatinine ≤ 1.6 mg/dl; alanine transaminase (ALT) and aspartate aminotransferase (AST) ≤ 3 times the normal range and total bilirubin ≤ 2.0 mg/dl; Pulmonary function ≤ grade 1 dyspnea (CTCAE v5.0) with oxygen saturation > 91% without oxygenation.
* subjects aged 15-65 years (including 15 and 65 years), regardless of gender.
* T-cell amplification test pass.
* expected survival > 3 months.

Exclusion Criteria:

* patients with recurrence of only isolated extramedullary lesions. combination of other malignant tumors.
* previously treated with anti-CD19 therapies.
* immunosuppressants use within 2 weeks prior to signing informed consent or plan to immunosuppressants after signing informed consent.
* uncontrolled active infections.
* HIV infection.
* active hepatitis B or hepatitis C infection.
* history of severe tachyphylaxis to aminoglycoside antibiotics.
* history or presence of clinically relevant Central Nervous System (CNS) pathology, such as epilepsy, generalized seizure disorder, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2030-04-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival（OS） | 4 years
  It is measured from the date of entry into this trial to the date of death from any cause; patients not known to have died at last follow-up are censored on the date they were last known to be alive.
leukemia free survival（LFS） | 4 years
  It is measured from the date of achievement of a remission until the date of relapse from CR, or CRi, or death from any cause; patients not known to have any of these events are censored on the date they were last examined.

SECONDARY OUTCOMES:
Number of adverse events | 4 years
  Adverse events are evaluated with CTCAE V5.0 from the date of entry into this trial.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No